CLINICAL TRIAL: NCT02632721
Title: An Open-label, Phase I/II Trial to Determine the Maximum Tolerated Dose and Investigate Safety, Pharmacokinetics and Efficacy of BI 836858 in Combination With Decitabine in Patients With Acute Myeloid Leukemia
Brief Title: A Trial to Find and Investigate a Safe Dose of BI 836858 in Combination With Decitabine for Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1315.2; 2015-002892-30 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; BI 836858

STUDY DESIGN:
Intervention Model Description: Phase I Dose Escalation: Open-label, single-arm, dose escalation
  - To determine the maximum tolerated dose (MTD) and the recommended dose for Phase I Extension (RExP1D)
  Phase I Extension: Open-label, two consecutive groups (cohort A and B) - To collect additional data on safety, pharmacokinetics and efficacy and to decide if the RExP1D will become the Recommended Phase II Dose (RP2D)
  Phase II: Open-label, two-arm randomized
  - To investigate efficacy, safety and pharmacokinetics of BI 836858 in combination with decitabine compared to decitabine monotherapy
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase I dose escalation: BI 836858 20 mg + decitabine (intensive) (Experimental): Dose escalation.
  Interventions: Drug: Decitabine; Drug: BI 836858
- Phase I dose escalation: BI 836858 40 mg + decitabine (intensive) (Experimental): Dose escalation.
  Interventions: Drug: Decitabine; Drug: BI 836858
- Phase I dose escalation: BI 836858 80 mg + decitabine (intensive) (Experimental): Dose escalation.
  Interventions: Drug: Decitabine; Drug: BI 836858
- Phase I Extension A: BI 836858 80 mg + decitabine (intensive) (Experimental): Extension phase.
  Interventions: Drug: Decitabine; Drug: BI 836858
- Phase I Extension B: BI 836858 80 mg + decitabine (standard) (Experimental): Extension phase.
  Interventions: Drug: Decitabine; Drug: BI 836858

INTERVENTIONS:
Drug: Decitabine
Drug: BI 836858

SUMMARY:
Phase I Dose Escalation:

Primary objective is to determine the Maximum Tolerated Dose (MTD) and the recommended dose for Phase I Extension.

Secondary objective is to investigate the safety, pharmacokinetics and efficacy of BI 836858 in combination with decitabine

Phase I Extension:

Primary objective is to collect additional data on safety, pharmacokinetics and efficacy and to define the Recommended Phase II Dose (RP2D) of BI 836858 in combination with decitabine.

Phase II: Primary objective is to investigate efficacy, safety and pharmacokinetics of BI 836858 in combination with decitabine compared to decitabine monotherapy.

ELIGIBILITY:
Inclusion criteria:

1)

Phase I Dose Escalation:

* Male or female patients >/= 18 years of age with relapsed or refractory AML
* Male or female patients >/= 65 years of age with previously untreated AML ineligible for receiving standard intensive therapy

Phase I Extension and Phase II:

-- Male or female patients >/= 65 years of age with previously untreated AML ineligible for receiving standard intensive therapy

2) Histologically or cytologically confirmed AML according to the WHO classification 3) Patients must be eligible for treatment with decitabine 4) Eastern co-operative oncology group (ECOG) performance score </=2 at screening Further inclusion criteria apply.

Exclusion criteria:

1. Acute promyelocytic leukemia (APL, French-American-British (FAB) subtype M3), according to WHO classification.
2. Patients who are candidates for allogeneic stem cell transplantation.
3. Active chronic graft versus host disease requiring immunosuppressive treatment.
4. Phase I extension and Phase II only:

   Prior treatment with a hypomethylating agent, such as prior treatment for Myelodysplastic Syndrome (MDS).
5. Prior treatment with Cluster of differentiation 33 (CD33) antibody. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (14):
- United States (4):
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Northwell Health, Lake Success, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
- Germany (6):
  - Universitätsklinikum Augsburg, Augsburg
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Münster, Münster
- A.O. Spedali Civili di Brescia, Brescia, Italy
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, Phase I/II trial to determine the maximum tolerated dose and investigate safety, pharmacokinetics and efficacy of BI 836858 in combination with decitabine in patients with acute myeloid leukemia.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive): 20 milligram (mg) of concentrate for solution for infusion of BI 836858 were administered as single dose via rate-controlled intravenous infusion once per week in 28-day treatment cycle (i.e. on Days 1, 8, 15, and 22 of the 28-day treatment cycles), together with 20 mg/square meter (m2) body surface area (BSA) of decitabine administered daily via intravenous infusion for 10 consecutive days (intensive treatment) from Day 1 to 10 in each treatment cycle. The BI 836858 dose was diluted in 0.9% sodium chloride to have full volume of the diluted compound 250 milliliter (mL).
- Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive): 40 milligram (mg) of concentrate for solution for infusion of BI 836858 were administered as single dose via rate-controlled intravenous infusion once per week in 28-day treatment cycle (i.e. on Days 1, 8, 15, and 22 of the 28-day treatment cycles), together with 20 mg/square meter (m2) body surface area (BSA) of decitabine administered daily via intravenous infusion for 10 consecutive days (intensive treatment) from Day 1 to 10 in each treatment cycle. The BI 836858 dose was diluted in 0.9% sodium chloride to have full volume of the diluted compound 250 milliliter (mL).
- Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive); Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive): 80 milligram (mg) of concentrate for solution for infusion of BI 836858 were administered as single dose via rate-controlled intravenous infusion once per week in 28-day treatment cycle (i.e. on Days 1, 8, 15, and 22 of the 28-day treatment cycles), together with 20 mg/square meter (m2) body surface area (BSA) of decitabine administered daily via intravenous infusion for 10 consecutive days (intensive treatment) from Day 1 to 10 in each treatment cycle. The BI 836858 dose was diluted in 0.9% sodium chloride to have full volume of the diluted compound 250 milliliter (mL).
- Phase I Extension B: BI 836858 80 mg + Decitabine (Standard): 80 milligram (mg) of concentrate for solution for infusion of BI 836858 were administered as single dose via rate-controlled intravenous infusion once per week in 28-day treatment cycle (i.e. on Days 1, 8, 15, and 22 of the 28-day treatment cycles), together with 20 mg/square meter (m2) body surface area (BSA) of decitabine administered daily via intravenous infusion for 5 consecutive days (standard treatment) from Day 1 to 5 in each treatment cycle. The BI 836858 dose was diluted in 0.9% sodium chloride to have full volume of the diluted compound 250 milliliter (mL).
Period: Overall Study
Arm/Group | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard)
Started | 4 | 3 | 9 | 15 | 18
Completed | 0 | 0 | 0 | 1 | 2
Not Completed | 4 | 3 | 9 | 14 | 16
Not completed — Adverse Event | 0 | 0 | 2 | 5 | 3
Not completed — Dose limiting toxicity | 0 | 0 | 0 | 1 | 0
Not completed — Progressive disease | 3 | 0 | 4 | 6 | 5
Not completed — Refused to continue taking trial medication | 0 | 1 | 1 | 1 | 2
Not completed — Inadequate clinical condition | 0 | 0 | 0 | 0 | 1
Not completed — No meet eligibility | 0 | 0 | 0 | 0 | 1
Not completed — Allergic reaction | 0 | 0 | 0 | 1 | 0
Not completed — Receiving Decitabine locally | 0 | 0 | 1 | 0 | 0
Not completed — No benefit from study treatment | 1 | 1 | 0 | 0 | 1
Not completed — Patient wish for other treatment | 0 | 1 | 0 | 0 | 0
Not completed — Relapsed Pneumonia | 0 | 0 | 0 | 0 | 1
Not completed — Therapy refractory AML | 0 | 0 | 0 | 0 | 1
Not completed — Increase of white blood cell count | 0 | 0 | 0 | 0 | 1
Not completed — Allogeneic peripheral blood stem cell transplantation | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: The treated set includes all patients who have received at least one dose of study medication (BI 836858 and/or decitabine).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard) | Total
Number analyzed (Participants) | 4 | 3 | 9 | 15 | 18 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.0 (11.34) | 52.3 (27.61) | 66.3 (13.02) | 74.9 (6.62) | 76.6 (4.24) | 72.3 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 7 | 6 | 20
  Male | 3 | 1 | 5 | 8 | 12 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 9 | 15 | 18 | 49
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Patients With Dose Limiting Toxicity (DLT(s)) During First Treatment Cycle
Description: Number of patients with dose limiting toxicity (DLT(s)) for BI 836858 in combination with decitabine during first treatment cycle (Phase 1).
  DLT was defined as any non-disease-related non-haematological adverse event (AE) of Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher. Expected non-haematological disease-related AEs were not to be regarded as a DLT.
  These included complications resulting from haematological AEs such as:
  * Bleeding and complications from bleeding due to thrombocytopenia as defined by the Investigator,
  * Infection and complications from infections due to neutropenia as defined by the Investigator,
  * Constitutional symptoms due to anaemia as defined by the Investigator
Time Frame: Up to 28 days (first treatment cycle).
Population: Treated set: All subjects who were documented to have received at least one dose of trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard)
Number analyzed (Participants) | 4 | 3 | 9 | 15 | 18
Participants | 0 | 0 | 0 | 1 | 1
Statistical Analysis 1: Comparison: Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive); Bayesian logistic regression model (BLRM) with overdose control was used to determine the maximum tolerated dose (MTD), defined as highest dose with less than 25% risk of the true DLT rate being equal to or above 33%; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.081 — Posterior probability of the DLT rate lying in the interval [0.16, 0.33) (target dosing) is reported
Statistical Analysis 2: Comparison: Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive); [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.33, 1) = 0 — Posterior probability of the DLT rate lying in the interval [0.33,1) (overdosing) is reported
Statistical Analysis 3: Comparison: Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive); [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.028 — Posterior probability of the DLT rate lying in the interval [0.16, 0.33) (target dosing) is reported
Statistical Analysis 4: Comparison: Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive); [analysis description as in outcome 1, analysis 1]; Test type: Other; Posterior probability of the DLT rate ly = 0 — Posterior probability of the DLT rate lying in the interval [0.33,1) (overdosing) is reported
Statistical Analysis 5: Comparison: Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive); [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.16, 0.33) = 0.012 — Posterior probability of the DLT rate lying in the interval [0.16, 0.33) (target dosing) is reported
Statistical Analysis 6: Comparison: Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive); [analysis description as in outcome 1, analysis 1]; Test type: Other; Probability of DLT rate in [0.33, 1) = 0 — Posterior probability of the DLT rate lying in the interval [0.33,1) (overdosing) is reported

2. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of BI 836858 in Combination With Decitabine
Description: The Maximum tolerated dose (MTD) of BI 836858 in combination with decitabine was estimated after the dose escalation part of the trial obtaining on the basis of dose limiting toxicities (DLT(s)) observed during the first treatment cycle. However, for those patients who receive more than one cycle of the combination treatment, all adverse events that constitute a DLT will be considered for re-estimation of the MTD based on the Bayesian logistic regression model (BLRM). The MTD is defined as the highest dose of BI 836858 (in combination with decitabine) with less than 25% risk of the true DLT rate being above 33% during the MTD evaluation period.
Time Frame: From first drug administration until end of treatment, up to 941 days.
Population: Maximum Tolerated Dose (MTD) evaluable set: This analysis set includes all subjects who were entered, treated and completed first cycle of planned treatment or subjects received at least 2 doses of BI 836858 due to BI 836858-related toxicity but not replaced.
Measure: Number; unit: milligram
Groups:
- Phase I: BI 836858 + Decitabine: Comprises all dose cohorts during the Phase I dose escalation and extension parts. 20/40/80 milligram (mg) of BI 836858 were administered as single dose via rate-controlled intravenous infusion once per week in 28-day treatment cycle (i.e. on Days 1, 8, 15, and 22 of the 28-day treatment cycles), together with 20 mg/square meter (m2) body surface area (BSA) of decitabine administered daily via intravenous infusion for 10 consecutive days (intensive treatment) from Day 1 to 10 (standard treatment: 5 consecutive days from Day 1 to 5) in each treatment cycle. The BI 836858 dose was diluted in 0.9% sodium chloride to have full volume of the diluted compound 250 milliliter (mL).
Arm/Group | Phase I: BI 836858 + Decitabine
Number analyzed (Participants) | 35
milligram | NA — No formal MTD was determined due to no DLTs were reported during dose escalation and only 2 DLTs were observed in the extension phase.

3. Secondary Outcome: Phase 1: Number of Patients With Objective Response (CR + CRi)
Description: Number of patients with objective response (Complete remission (CR) + complete remission with incomplete remission (CRi)).
  CR was defined as bone marrow (BM) blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1.0 x 109/L [1,000/μL]; platelet count > 100 x 109/L [100,000/μL]; independence of red blood cells transfusions (no transfusion for 1 week prior to the assessment). No minimum duration of response is required.
  CRi was defined as all CR criteria except for residual neutropenia (< 1.0 x 109/L [1,000/μL]) or thrombocytopenia (< 100 x 109/L [100,000/μL]).
Time Frame: From start of treatment until the earliest of progression, death or end of trial, up to 971 days.
Population: Treated set: All subjects who were documented to have received at least one dose of trial medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard)
Number analyzed (Participants) | 4 | 3 | 9 | 15 | 18
Participants
  Objective response (CR + CRi) | 2 | 0 | 6 | 7 | 4
  Complete remission (CR) | 1 | 0 | 1 | 3 | 3
  Complete remission with incomplete recovery (CRi) | 1 | 0 | 5 | 4 | 1

ADVERSE EVENTS:
Time Frame: From first administration of trial medication until 30 days of residual effect period after the last administration of trial medication, up to 971 days.
Description: Treated set: All subjects who were documented to have received at least one dose of trial medication.
Arm/Group | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard)
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/3 | 5/9 | 11/15 | 13/18
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 8/9 | 14/15 | 17/18
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 9/9 | 15/15 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) (N=4) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) (N=3) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) (N=9) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) (N=15) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 5 | 5
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 3 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Cardiac valve abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 2 | 4
Sepsis (Infections and infestations) | 0 | 1 | 1 | 2 | 3
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2 | 5 | 5
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoglossal nerve paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation: BI 836858 20 mg + Decitabine (Intensive) (N=4) | Phase I Dose Escalation: BI 836858 40 mg + Decitabine (Intensive) (N=3) | Phase I Dose Escalation: BI 836858 80 mg + Decitabine (Intensive) (N=9) | Phase I Extension A: BI 836858 80 mg + Decitabine (Intensive) (N=15) | Phase I Extension B: BI 836858 80 mg + Decitabine (Standard) (N=18)
Acquired antithrombin III deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 6 | 4 | 6
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 1 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0
Eye haematoma (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eyelid bleeding (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 4 | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 6 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 0 | 5 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 2
Catheter site pain (General disorders) | 1 | 0 | 1 | 0 | 0
Catheter site thrombosis (General disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 2 | 2 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 3 | 2 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 2 | 2
Implant site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 1 | 1 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 3 | 3 | 4
Oedema peripheral (General disorders) | 2 | 1 | 4 | 7 | 6
Pain (General disorders) | 1 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 1 | 2 | 4 | 4
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Treatment noncompliance (General disorders) | 0 | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Vessel puncture site swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cerebral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1
Ecthyma (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 1 | 1 | 2 | 1
Herpes simplex viraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 1 | 0 | 0 | 2
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 3
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3 | 4 | 8 | 11
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Transplantation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 2
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 2 | 1 | 1
Cortisol decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 3 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 2 | 2
Platelet count decreased (Investigations) | 1 | 2 | 4 | 3 | 5
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 1
Prothrombin time shortened (Investigations) | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 2 | 3 | 2 | 5
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 3 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 3 | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 4 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoglossal nerve paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 2 | 2 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 1 | 3
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 4 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 3 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 3 | 0 | 1 | 2 | 3
Hypertension (Vascular disorders) | 3 | 2 | 3 | 4 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 2 | 2
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Illness (General disorders) | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Sponsor stopped development of the study drug before Phase II start. Phase II was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02632721/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT02632721/SAP_001.pdf